CLINICAL TRIAL: NCT06067386
Title: Selective Reporting for Antibiotic Susceptibility Testing and GPs' Prescribing of Broad-spectrum Antibiotics in Women With E. Coli UTIs
Acronym: ABC-MG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RC22_0003
Record Dates: First submitted 2023-09-22; First posted 2023-10-04 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-09

CONDITIONS: Urinary Tract Infections
Keywords: Antibiotic therapy; General practice; Primary care; Public health
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): For each E. coli positive urine culture analyzed by LabOuest, GPs will receive an antibiotic susceptibility testing report, with the list of antibiotics restricted according to four E. coli susceptibility profiles, with an emphasis on narrower-spectrum antibiotics. The selected antibiotic susceptibility testing was developed following a targeted literature review and consultation with a steering committee including GPs, biologists and infectiologists. At the GP's request, a full antibiogram can be provided.
  Interventions: Other: Dissemination of a selective reporting for antibiotic susceptibility testing
- Control arm (Active Comparator): GPs will receive a standard antibiotic susceptibility testing report for each E. coli positive urine culture.
  Interventions: Other: Standard antibiotic susceptibility testing report

INTERVENTIONS:
Other: Dissemination of a selective reporting for antibiotic susceptibility testing — For each E. coli positive urine culture analyzed by LabOuest, GPs will receive an antibiotic susceptibility testing report, with the list of antibiotics restricted according to four E. coli susceptibility profiles, with an emphasis on narrower-spectrum antibiotics. The selected antibiotic susceptibility testing was developed following a targeted literature review and consultation with a steering committee including GPs, biologists and infectiologists. At the GP's request, a full antibiogram can be provided.
  Arms: Intervention arm
Other: Standard antibiotic susceptibility testing report — GPs will receive a standard antibiotic susceptibility testing report for each E. coli positive urine culture.
  Arms: Control arm

SUMMARY:
The control of antibiotic resistance requires a reduction in inappropriate prescriptions of broad-spectrum antibiotics (amoxillin-clavulanate (AMC), fluoroquinolones (FQ), third-generation cephalosporins (C3G)), particularly for urinary tract infections treated in primary care. Several studies have reported the positive impact of antibiotic susceptibility testing performed on urine cultures on the appropriate use of antibiotics.

The "selective reporting for antibiotic susceptibility testing ", defined as the restriction of the list of antibiotics mentioned in the report according to the antibiotic resistance profile, would allow, according to observational studies, a reduction of 25 to 70% of the initial prescriptions of broad-spectrum antibiotics and a 20% rate of antibiotic de-escalation (=reduction of the antibacterial spectrum of an antibiotic treatment after re-evaluation).

The objective is to assess the impact of disseminating a selective reporting for antibiotic susceptibility testing on the dispensing of broad-spectrum antibiotics prescribed by general practitioners (GPs) for E. coli positive urine cultures in adult women, compared to the dissemination of a standard antibiotic susceptibility testing.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* women ≥18 years of age,
* affiliated with the CPAM of Loire Atlantique (44) or Maine et Loire (49),
* with a urine culture: i) analyzed by LabOuest, ii) positive for E. coli, and iii) associated with a prescription for antibiotics by a general practitioner in the period 7 days before and 14 days after the antibiotic susceptibility testing.

General practitioners :

* practicing in primary care Loire Atlantique (44) and/or Maine et Loire (49),
* having been consulted by at least 100 different patients in the 12 months prior to baseline,
* having received at least one urine culture result for a woman ≥18 years of age analyzed by LabOuest over the 12 months prior to baseline.

Exclusion Criteria:

Patients :

* hospitalized in the period 7 days before and 14 days after antibiotic susceptibility testing (data on antibiotics dispensed in healthcare institutions are not accessible via DCIR data),
* with reimbursements for antibiotics prescribed by physicians in different practices over the period 7 days before and 14 days after antibiotic susceptibility testing.

General practitioners :

* with a special practice (acupuncture, allergology, angiology).
* not receiving any urine culture results analyzed by a laboratory of the LabOuest network in the year following the intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-11-21 (Estimated); Study Completion 2024-11-21 (Estimated)

PRIMARY OUTCOMES:
Rate of broad-spectrum antibiotic dispensing | 5 days
  The primary endpoint will be the rate of broad-spectrum antibiotic dispensing, defined as the number of urine cultures associated with a prescription of broad-spectrum antibiotics (Amoxicillin/clavulanic acid, fluoroquinolone, third-generation cephalosporin) prescribed by GPs in the same practice over a period from 3 days before to 5 days after report of the antibiotic susceptibility testing, relative to the total number of urine cultures. This period of interest corresponds to the period of empirical antibiotic therapy (=within 3 days before report of the antibiotic susceptibility testing), and the period of directed antibiotic therapy (=within 5 days after report of the antibiotic susceptibility testing).
  A sensitivity analysis of the primary endpoint will be carried out by varying the time window for broad-spectrum antibiotic dispensing around the date of the antibiotic susceptibility testing result, up to a maximum of 7 days before and 14 days after.

SECONDARY OUTCOMES:
Rate of directed broad-spectrum antibiotic dispensing (=within 5 days after report of the antibiotic susceptibility testing) | 5 days
  This analysis will be restricted to women who have received no empirical antibiotic therapy (=within 3 days before report of the antibiotic susceptibility testing)
"Antibiotic de-escalation" rate: modification of an empirical broad-spectrum antibiotic therapy to a directed narrow-spectrum antibiotic therapy | 5 days
Rate of broad-spectrum antibiotic dispensing as a function of the number of selective antibiotic susceptibility testings received per practice, as a continuous variable ("dose-effect") and ordinal variable ("threshold-effect") | 5 days
GP characteristics: demographics (age, gender), practice patterns (type of practice commune based on INSEE urban area zoning), number of encounters/year, and number of patients declared | 5 days
  Impact of targeted antibiotic susceptibility testing compared to of a standard antibiotic susceptibility test as a function of GP characteristics
Patient characteristics (age, diabetes, pregnancy, nursing home) | 5 days
  Impact of targeted antibiotic susceptibility testing compared to of a standard antibiotic susceptibility test according to patient characteristics,
E.coli antimicrobial susceptibility profiles | 5 days
  Impact of targeted antibiotic susceptibility testing compared to of a standard antibiotic susceptibility test based on E. coli antimicrobial susceptibility profiles

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France